CLINICAL TRIAL: NCT06572813
Title: Bortezomib Combined with PD-1 MAb and MFOLFIRINOX for First-line Treatment of Metastatic Pancreatic Cancer：An Exploratory Clinical Trial
Brief Title: Bortezomib Combined with PD-1 MAb and MFOLFIRINOX for Metastatic Pancreatic Cancer
Acronym: CISPD-7
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CISPD-7
Record Dates: First submitted 2024-08-21; First posted 2024-08-27 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-08

CONDITIONS: Pancreas Cancer
Keywords: metastatic pancreatic cancer; bortezomib; PD-1 antibody; chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bortezomib; sintilimab

STUDY DESIGN:
Intervention Model Description: Phase 1 (Evaluation of Drug Tolerance) Primary objective: To evaluate the tolerability of bortezomib, PD-1 mAb and mFOLFIRINOX in patients with advanced metastatic pancreatic cancer, and to determine the dose of bortezomib in the combination regimen; Secondary objectives: To evaluate the immunogenicity characteristics and safety of the combination regimen of bortezomib, PD-1 mAb and mFOLFIRINOX in patients with advanced metastatic pancreatic cancer; Phase 2 (Dose Expansion) Primary objective: To evaluate the tolerability and efficacy of the combination regimen of bortezomib, PD-1 mAb and mFOLFIRINOX in subjects with advanced metastatic pancreatic cancer; Secondary Objective: To evaluate the immunogenicity and safety of bortezomib, PD-1 mAb and mFOLFIRINOX in subjects with advanced metastatic pancreatic cancer; and to explore biomarkers related to combination therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1 (Drug Tolerance Evaluation) (Experimental): Using a 3 + 3 trial design, bortezomib dose exploration was performed to determine the stage 2 bortezomib dose. The number of participants at this stage is 6-9.
  Interventions: Drug: Bortezomib Injection; Drug: Sintilimab; Drug: mFOLFIRINOX
- Phase 2 (Dose extension) (Experimental): Phase 2: This phase will adopt competitive enrollment, and the Bayesian prediction probability method will be used to monitor the main efficacy index of the trial ORR in real time to determine the early termination or continue the trial. A maximum number of 57 patients were enrolled in this stage.
  Interventions: Drug: Bortezomib Injection; Drug: Sintilimab; Drug: mFOLFIRINOX

INTERVENTIONS:
Drug: Bortezomib Injection — Bortezomib Injection, a kind of chemotherapy drug
Drug: Sintilimab — PD-1 antibody
Drug: mFOLFIRINOX — Combination of oxaliplatin, fluorouracil, irinotecan, leucovorin calcium

SUMMARY:
This is an single-center, prospective, open-label clinical trial, to explore the safty and efficacy of combination of Bortezomib, Sindilizumab, and mFOLFIRINOX Chemotherapy (oxaliplatin, fluorouracil, irinotecan, leucovorin) in metastatic pancreatic cancer

DETAILED DESCRIPTION:
Phase 1 (Evaluation of Drug Tolerance) Primary objective: To evaluate the tolerability of bortezomib, PD-1 mAb and mFOLFIRINOX in patients with advanced metastatic pancreatic cancer, and to determine the dose of bortezomib in the combination regimen; Secondary objectives: To evaluate the immunogenicity characteristics and safety of the combination regimen of bortezomib, PD-1 mAb and mFOLFIRINOX in patients with advanced metastatic pancreatic cancer; Phase 2 (Dose Expansion) Primary objective: To evaluate the tolerability and efficacy of the combination regimen of bortezomib, PD-1 mAb and mFOLFIRINOX in patients with advanced metastatic pancreatic cancer; Secondary Objective: ORR; PFS; OS; and to evaluate the immunogenicity and safety of bortezomib, PD-1 mAb and mFOLFIRINOX in subjects with advanced metastatic pancreatic cancer; and to explore biomarkers related to combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) confirmed pancreatic ductal adenocarcinoma (PDAC).
* Recurrent disease or metastatic disease (such as liver, peritoneum, lung) evaluated by abdominal contrast-enhanced CT, MRI, and chest CT. PET/CT or other imaging examinations would be used if necessary.
* Never receive any systematic treatment or Progression after fisrt line Gemcitabine base chemotherapy
* ECOG score 0 or 1.
* Serum creatinine level is normal, and serum total bilirubin level is less than 1.5 x ULN.
* ALT and AST are less than 2 x ULN.
* Signed informed consent.

Exclusion Criteria:

* History of participation of other clinical trails within 4 weeks
* History of autoimmune disease or other condition receiving glucocorticoid treatment
* History of receiving chemotherapy within 2 weeks
* History of radiotherapy and molecular target therapy within 2 weeks
* History if active tuberculosis
* History of malignance treatment in the past, excluding basal and cutaneous squamous cell carcinoma, cervical carcinoma in situ, papillary thyroid carcinoma
* Major cardiovascular diseases (including myocardial infarction, unstable angina, congestive heart failure, severe uncontrolled arrhythmia) during the past six months of enrollment.
* Hematological precancerous diseases, such as myelodysplastic syndromes.
* Evidence of clinical-related or previous interstitial lung disease, such as noninfectious pneumonia or pulmonary fibrosis, or baseline chest CT scan or chest X-ray findings
* Previous or physical findings of central nervous system disease, except for adequately treated (e.g. primary brain tumors, uncontrolled seizures or strokes with standard medications)
* Preexisting neuropathy > 1 (NCI CTCAE).
* Immune deficiency syndrome, such as active tuberculosis and HIV infection.
* Allograft requires immunosuppressive therapy or other major immunosuppressive therapies.
* Severe serious wounds, ulcers or fractures.
* Clinical evaluation is unacceptable

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to 2 years.
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0，including Complete Blood Count, liver function, renal function lab test and other blood test will be evaluated by using CTCAE 5.0 during study.
Phase 2: Objective reponse rate (ORR) | Up to 2 years
  The proportion of patients who had tumor evaluated as PR according to RECIST1.1 criteria during phase 2

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to 2 years
  The proportion of patients who had tumor evaluated as PR or SD according to RECIST1.1 criteria during phase 2
Duration of remission （DoR） | Up to 2 years
  The time from the first assessment of the tumor as CR or PR to the first assessment of PD or death from any cause during phase 2
Progression-free survival （PFS） | Up to 2 years
  The time from enrolled to disease pregression or death from any cause during phase 2
Overall survival (OS) | Up to 2 years
  The time from enrolled to death from any cause during phase 2

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Liang, Principal Investigator — Zhejiang University
Locations (1):
- First Affiliated Hospital of Zhejiang University Schlool of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No